CLINICAL TRIAL: NCT01397604
Title: A Randomized, Blinded, Placebo-Controlled Phase 1 Study to Evaluate the Safety and Immunogenicity of GLA in Healthy Volunteers
Brief Title: The Effects of GLA on Human Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: IDRI Corporation (Unknown); Immune Design, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BYI-0736
Record Dates: First submitted 2011-07-14; First posted 2011-07-19 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — GLA-AF adjuvant; glucopyranosyl lipid-A; Squalene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Saline Placebo (No Intervention): The trial will consist of a total of 32 people. An over-enrollment of about 10% (3 volunteers) will be permitted.
  Each cohort will be recruited in sequence. Cohort I will include 16 subjects that will receive a subcutaneous injection, randomized equally so that 5 individuals will receive GLA-AF (2µg), 5 individuals will receive GLA-SE, 3 individuals will receive saline placebo and 3 individuals will receive SE vehicle. Cohort II will include 16 subjects that will receive intramuscular injections, randomized equally into 5 GLA-AF (2µg) subjects, 5 GLA-SE (2µg) subjects, 3 saline placebo subjects and 3 SE vehicle control subjects.
- SE Vehicle (Placebo Comparator): The trial will consist of a total of 32 people. An over-enrollment of about 10% (3 volunteers) will be permitted.
  Each cohort will be recruited in sequence. Cohort I will include 16 subjects that will receive a subcutaneous injection, randomized equally so that 5 individuals will receive GLA-AF (2µg), 5 individuals will receive GLA-SE, 3 individuals will receive saline placebo and 3 individuals will receive SE vehicle. Cohort II will include 16 subjects that will receive intramuscular injections, randomized equally into 5 GLA-AF (2µg) subjects, 5 GLA-SE (2µg) subjects, 3 saline placebo subjects and 3 SE vehicle control subjects.
  The SE (squalene) vehicle contains the oil emulsion in which the GLA-SE is solubilized.
  Interventions: Other: Squalene
- GLA-AF (Active Comparator): The trial will consist of a total of 32 people. An over-enrollment of about 10% (3 volunteers) will be permitted.
  Each cohort will be recruited in sequence. Cohort I will include 16 subjects that will receive a subcutaneous injection, randomized equally so that 5 individuals will receive GLA-AF (2µg), 5 individuals will receive GLA-SE, 3 individuals will receive saline placebo and 3 individuals will receive SE vehicle. Cohort II will include 16 subjects that will receive intramuscular injections, randomized equally into 5 GLA-AF (2µg) subjects, 5 GLA-SE (2µg) subjects, 3 saline placebo subjects and 3 SE vehicle control subjects.
  GLA-AF contains the study drug in an aqueous solution.
  Interventions: Drug: GLA-AF
- GLA-SE (Active Comparator): The trial will consist of a total of 32 people. An over-enrollment of about 10% (3 volunteers) will be permitted.
  Each cohort will be recruited in sequence. Cohort I will include 16 subjects that will receive a subcutaneous injection, randomized equally so that 5 individuals will receive GLA-AF (2µg), 5 individuals will receive GLA-SE, 3 individuals will receive saline placebo and 3 individuals will receive SE vehicle. Cohort II will include 16 subjects that will receive intramuscular injections, randomized equally into 5 GLA-AF (2µg) subjects, 5 GLA-SE (2µg) subjects, 3 saline placebo subjects and 3 SE vehicle control subjects.
  GLA-SE contains the study drug in a squalene oil emulsion.
  Interventions: Drug: GLA-SE

INTERVENTIONS:
Drug: GLA-AF — GLA-AF contains GLA, a new synthetic lipid A molecule that combines 6 acyl chains with a single phosphorylation site. GLA-AF contains GLA in an aqueous solution. One 2 mcg injection will be given per patient in the upper arm, each randomized to either subcutaneous or intramuscular routes.
  Arms: GLA-AF
Drug: GLA-SE — GLA-SE contains GLA, a new synthetic lipid A molecule that combines 6 acyl chains with a single phosphorylation site. GLA-SE contains GLA in a squalene oil emulsion. One 2 mcg injection will be given per patient in the upper arm, each randomized to either subcutaneous or intramuscular routes.
  Arms: GLA-SE
Other: Squalene — Squalene is a natural organic compound obtained from shark liver oil. In this study, it is used to solubilize GLA in the GLA-SE formulation. Patients randomized to receive the squalene will be given one 2mcg injection of the squalene oil in the upper arm, each patient randomized further to either subcutaneous or intramuscular routes.
  Arms: SE Vehicle

SUMMARY:
The advent of vaccines contributed to major improvements in human morbidity and mortality due to infectious diseases such as polio, small pox, measles and diphtheria. However infectious diseases like HIV, malaria and tuberculosis continue to be major causes of death worldwide and conventional vaccine strategies have not been successful. The fundamental problem is that current protein based vaccines do not elicit the necessary T-cell immunity. Experimentally, adjuvants can be given in conjunction with a vaccine to activate and mature the dendritic cell (DC), which can then direct an immune response to enhance T-cell immunity. One family of potential adjuvants functions through the activation of Toll-like receptors (TLR) on the DC. Major gaps exist in our understanding of adjuvant effects in humans. We hypothesize that a synthetic adjuvant directed to activate TLR4 (GLA) will safely stimulate the innate immune system when administered subcutaneously (SC) or intramuscularly (IM). Importantly, in contrast to other adjuvant trials in which adjuvant is combined with an antigen or vaccine, GLA will be tested in isolation. This is because we anticipate the future administration of GLA with our dendritic cell targeted HIV vaccine. A DC-targeted vaccine cannot be given without an immune stimulating adjuvant due to potential risk of inducing immune tolerance. Therefore, in order to understand the specific contributions of GLA versus the DC-targeted vaccine, we need to understand the GLA effects in isolation. The safety and tolerability of 2 different formulations of GLA (GLA-SE vs. GLA-AF) administered by 3 different routes (SC, ID, IM) will be the major focus of this trial. The second focus will be characterizing the innate immune response by assessing systemic cytokine and chemokine levels and determining global gene regulation following GLA stimulation. The third focus will be on the cellular effects of GLA, specifically on blood monocytes and dendritic cells. Monocytes may represent a large pool of inducible potent DC (monocyte-derived DC), however these cells have not been well characterized in humans. We will investigate the effects of GLA stimulation on the peripheral blood monocyte subsets that might give rise to monocyte-derived DC.

DETAILED DESCRIPTION:
Vaccines against infectious diseases have been instrumental to the improvement of human health and remain a pillar of modern public health strategies. Yet serious life threatening infections including HIV, malaria and tuberculosis remain a global problem and pandemic diseases like influenza continue to threaten human life. As well, vaccines are now being pursued in the areas of cancer prevention and treatment. A fundamental barrier that has prevented effective vaccines for many diseases is that conventional protein based vaccines do not elicit the critical requirement of T-cell mediated immunity. One approach to generating an improved T-cell response to a vaccine has been to identify new protein target candidates. This approach has not resulted in significant advances in vaccine development. We are interested in a novel approach that combines specific immune stimulants, or adjuvants, with a vaccine target to optimize and enhance the desired T-cell immune response. The development and study of novel adjuvants like GLA will allow us to further our investigation into dendritic cell targeted vaccines leading to improved vaccines for many diverse diseases.

Toll-Like Receptor (TLR) Background The TLR's are type 1 transmembrane receptors that share a leucine-rich repeat domain (LRR) in the extracellular loop and a Toll/IL-1 receptor (TIR) homology domain in the intracellular tail. The importance of TLRs to host defense and immunity was first appreciated in Drosophila that became susceptible to fungal infections following genetic deletion of the toll genes. Mammalian homologs were identified soon after using a mouse strain that was well known to be highly susceptible to Gram-negative infections and were hyporesponsive to lipopolysaccharide (LPS). These mice were found to have a mutational change on the TLR4 gene, rendering it non-functional and this discovery solidified the existence and importance of the Toll proteins in mammals. Mice with genetic deletions of TLR4 demonstrated the importance of TLR to bacterial infections and provided clear evidence that TLR4 was specific for Gram negative infections. Currently 10 functional TLRs have been discovered in humans and extensive research has identified a number of pathogen-derived agonists for specific TLRs. It is generally accepted that the TLR's function by recognizing conserved structures of an organism or pathogen associated molecular patterns (PAMPs). Clearly these innate receptors are critical to surviving a microbial insult as they provide a first line of defense that is not dependent on generating a specific T-cell and B-cell response, a process that can take weeks. Despite their clear role in innate immunity, evidence is accumulating that TLR stimulation has potent influence on the development of T and B cell mediated immunity through the activation and maturation of dendritic cells (DC). This knowledge has led to the development of TLR-based vaccine adjuvants that activate and mature DC.

Monocyte and Dendritic Cell Overview Dendritic cells (DC) are part of the innate and adaptive immune systems and reside at host-microbial interfaces including the surfaces of the gut, lung and within the skin. These cells constantly survey their environment in search of microbial pathogens through the expression of several families of pattern recognition receptors (PRR) including the Toll-like receptors (TLR). Immature DC are particularly efficient in antigen uptake and processing, while activated DC mature and become potent antigen presenting cells to T-lymphocytes. Importantly, immature DC have the potential to induce immune tolerance by deleting antigen specific T cells, resulting in no immune response. Activated DC however direct the immune response through the release of particular cytokines. Different initial stimuli will influence DC to drive CD4+ T-cells to differentiate along very divergent functional pathways including Th1, Th2, Th17 and Treg. Therefore, DC are critical to appropriate innate host defense as well as to orchestrate an adaptive response. Given their pivotal role in host defense, DC are relatively rare cells that, at steady state, develop independently from other blood cells. Enhancing and directing the function and quantity of DC will provide benefit to both host defenses as well as to vaccine science. The Steinman lab has pioneered a novel method of vaccination by targeting the antigen of interest specifically to the DC population. DC-targeted vaccines have shown promise in animal models and a DC-targeted HIV vaccine has recently been administered to humans for the first time.

Monocytes are a more abundant cell type that account for approximately 10% of blood leukocytes in humans and 4% in mice. Monocytes are peripheral blood effector cells that participate in host defense and are efficient scavenging cells. They serve as precursors to tissue macrophages. In humans, 3 subsets of monocytes have been proposed based on cell surface expression of CD14 and CD16, while 2 subsets exist in mice and are marked by CD115 and Ly6C. The role of these subsets during innate immunity requires further investigation. Evidence suggests that monocytes can be induced to differentiate into DC, however definitive in vivo evidence of this was previously lacking. Recent work in the Steinman lab has shown that in vivo authentic DC can be rapidly differentiated and mobilized from the larger monocyte pool in times of acute inflammation and infection. This rapid re-deployment could be induced by either gram-negative bacteria or LPS and was entirely dependent on TLR4. Similarly, human monocytes can de induced to differentiate into DC, however the understanding of this process is limited to in vitro cell culture with large gaps in our understanding of in vivo human monocyte derived-DC. Preliminary data suggests that GLA administration in mice, like LPS, can mobilize the monocyte pool into becoming Mo-DC. It is unknown if human monocytes in vivo rapidly expand the DC population following administration of TLR4 adjuvant GLA. Understanding the mechanisms of this re-deployment will further our understanding of how to rapidly expand and harness the utility of DC using adjuvants. Ultimately, we anticipate that adjuvant-specific DC responses will improve T-cell immunity and enhance vaccine effectiveness.

Rationale for Investigating an Adjuvant in Isolation The standard adjuvant trial consists of the adjuvant under investigation combined with a known licensed vaccine but not in isolation. However, as previously described, we are hopeful that GLA may become an important adjuvant of our DC-targeted HIV vaccine currently in development. The DC represents the most potent antigen-presenting cell and specifically targeting an antigen of interest to this cell generates improved immune responses. However there are important considerations when targeting antigen to DC. Immature unstimulated DC that encounter an antigen have the ability to delete antigen specific T cells thereby causing tolerance and a DC-targeted antigen vaccine alone may cause immune tolerance. In contrast DC that have matured are able to induce potent effector T cell responses to the targeted antigen. DC can be activated by TLR stimulation and therefore combining TLR stimulated DC maturation with a DC-targeted antigen would result in optimal T cell mediated immunity. In theory the DC-targeted vaccine could never be given without a DC maturing adjuvant and the specific effects and actions of GLA would not be known unless it was studied first in isolation. To plan an eventual DC-targeted HIV vaccine trial with an adjuvant, it will also be critical to know the temporal immune effects of isolated GLA.

GLA Background Information GLA is a new completely synthetic lipid A (active component of natural LPS) molecule that combines 6 acyl chains with a single phosphorylation site. The advantage of this LPS-like molecule is that it is not purified from a bacterial source thereby allowing a homogenous solution only containing molecules with 6 acyl chains. This is important because 6 acyl chains results in maximal TLR4 activation while lipid A molecules with 5 or 7 acyl chains are 100 times less active and 4 acyl chains is immuno-inhibitory. MPL is an existing TLR4 vaccine adjuvant that is derived from salmonella LPS and represents a heterogeneous mixture of 3, 4, 5 and 6 acylated molecules. MPL induces effective humoral antibody response during vaccination, but it does not generate CD4 T-cell immunity, making it an undesirable adjuvant for many protein-based vaccines. In animal models GLA added to the Fluzone vaccine improves humoral and cellular immunity to influenza. GLA has been tested in humans for safety in combination with an influenza vaccine however its individual effects have not been studied. Particularly the isolated effects on cytokine, chemokine and gene regulation in humans is not known and monocytes subsets were not previously investigated.

The optimal formulation and route of administration are not known; therefore a major component of this investigation will be to determine a safe and tolerable formulation and route. GLA has been administered to humans in combination with the Fluzone vaccine ranging in doses from 0.5μg to 5μg intramuscularly; however it has not been tested in isolation, and only the oil-in-water stable emulsion (GLA-SE) was used. Fluzone is a reactogenic vaccine and dose-limiting toxicity did occur in 3 of 4 patients who received Fluzone + high dose GLA-SE (5μg), but a good safety profile was observed between 0.5-2.5μg. The stable emulsion (SE) contains squalene and was used at 2% (vol:vol). We will continue to use this percentage in our GLA-SE formulation. A second formulation of GLA has subsequently been developed to avoid the need for an emulsion; GLA-AF is aqueous and should theoretically have a reduced side-effect profile and less reactogenicity than GLA-SE. We plan to compare the two formulations of GLA in isolation; GLA-SE (stable emulsion) and GLA-AF (aqueous formulation). GLA-AF has never been administered to humans and therefore this version represents a first-in-human trial. For safety reasons GLA-AF injections must be separated by a day and since it will not be possible to know who will receive GLA-AF, we will inject the first nine subjects in each cohort one day apart. Due to the complexity of the number of groups in this study, we will enroll and complete each route sequentially as a cohort. The subcutaneous cohort will be the first group screened, enrolled, randomized and injected, followed by intramuscular.

Summary This study will be a phase-1, randomized, placebo-controlled, double-blinded clinical trial to compare GLA formulation and administration route in humans. Safety and tolerability of the different formulations (GLA-SE vs. GLA-AF) and routes (SC, IM, ID) will be the primary focus. Our second focus will be to detail the global immune response be measuring systemic cytokines, chemokines and global gene regulation. The third focus will be to investigate the effects of GLA on the peripheral blood immune cells including monocytes and dendritic cells. This study will add first-in-human data on GLA-AF and detail the isolated effects of GLA on the innate immune system. The results of this trial will lay the foundation for a true adjuvant trial using GLA + antigen and ultimately to use GLA to adjuvant our DC-targeted vaccine in humans.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males and females, as assessed by a medical history, physical exam, and laboratory tests
2. Age of at least 18 years of age on the day of screening and no greater than 60 years at time of administration
3. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study (screening plus 4 weeks)
4. Willing to undergo HIV testing and counseling and receive HIV test results
5. If a female of child bearing potential, must be willing to use two effective methods of contraception (combined oral contraceptive pill; injectable contraceptive; diaphragm; Intra Uterine Device (IUD); condoms; anatomical sterility in self or partner) throughout until 6 weeks after study drug administration. If a sexually active male, must be willing to use two effective methods of contraception (such as condoms, anatomical sterility) from screening until 6 weeks after study drug administration (same as above) and will be advised not to get his partner(s) pregnant during this time.

Exclusion Criteria:

1. Confirmed HIV-1 or HIV-2 infection
2. Any clinically significant abnormality on medical history or physical examination including history of immunodeficiency or autoimmune disease
3. Any use of systemic corticosteroids immunosuppressive anticancer medications
4. Any clinically significant acute or chronic medical condition requiring care of a physician (e.g., diabetes, coronary artery disease, rheumatologic illness, malignancy, substance abuse) that in the opinion of the investigator would preclude participation
5. Any laboratory value outside of reference range other than CRP, with the exception of any non-clinically significant Grade I elevations of liver function tests (AST, ALT, direct/total bilirubin), electrolytes (Na, K, Cl, CO2), CBC, urinalysis as determined by the Principal Investigator or his designee.
6. Within the 12 months prior to enrollment, the subject self reports excessive daily alcohol use, frequent binge drinking or chronic marijuana abuse (defined as greater than 2 times a week) or any other use of illicit drugs
7. Positive hepatitis B surface antigen, positive hepatitis C antibodies, or active syphilis infection based on clinical evaluation;
8. If female, pregnant, planning a pregnancy during the trial period, or lactating
9. Receipt of a live attenuated vaccine within 30 days or other vaccine within 14 days prior to study drug
10. Participation in another clinical study of an investigational product currently or within past 12 weeks, or expected participation during this study
11. In the opinion of the investigator, unlikely to comply with protocol due to medical, social or psychiatric reasons
12. Allergy to eggs
13. A glomerular filtration rate that is less than 60mL/min/1.73 m2 as calculated by study team based on laboratory creatinine values.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 6 months
  Local reactogenicity events and systemic reactogenicity events will be monitored.
  Local reactogenicity events:Moderate significant events include, but are not limited to, pain, tenderness, erythema, skin discoloration, edema, vesicle formation or ulceration, induration, pruritus, and formation of a crust or scab.
  • Systemic reactogenicity events: Include fever, chills, headache, nausea, vomiting, malaise, myalgia, arthralgia, and rash.

SECONDARY OUTCOMES:
Global Innate Immune Responses | 1 year
  Serum will be analyzed for the expression of soluble immune molecules including cytokines and chemokines.
  Examining the expression of cell surface molecules using multicolor flow cytometry will assess peripheral monocyte subset activation and characterization.
  Whole blood global gene arrays will be used to assess GLA stimulated gene regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Caskey, MD, Principal Investigator — Instructor in Clinical Investigation
Locations (1):
- The Rockefeller University, New York, New York, United States